CLINICAL TRIAL: NCT04249167
Title: Cryoablation and Anti-PD-L1 Immunotherapy for Triple Negative Breast Cancer (TNBC)
Brief Title: Cryoablation, Atezolizumab/Nab-paclitaxel for Locally Advanced or Metastatic Triple Negative Breast Cancer
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: study was dropped
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC2031; NCI-2020-00333 (Other Grant/Funding Number: CTRP (Clinical Trial Reporting Program)); 19-008704 (Other: Mayo Clinic in Florida)
Record Dates: First submitted 2020-01-27; First posted 2020-01-30 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2021-12

CONDITIONS: Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Anatomic Stage IV Breast Cancer AJCC v8; Locally Advanced Breast Carcinoma; Metastatic Triple-Negative Breast Carcinoma; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8; Prognostic Stage IV Breast Cancer AJCC v8
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — atezolizumab; Cryosurgery; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Taxes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (cryoablation, atezolizumab, nab-paclitaxel) (Experimental): Patients undergo cryoablation of the primary tumor over about 1 hour. After 2-3 weeks, patients receive atezolizumab IV on days 1 and 15 and nab-paclitaxel IV on days 1, 8, and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Atezolizumab; Procedure: Cryosurgery; Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG7446; RO5541267; Tecentriq
Procedure: Cryosurgery — Undergo cryoablation of the primary tumor
  Other Names: Ablation, Cryo; Cryoablation; cryosurgical ablation
Drug: Nab-paclitaxel — Given IV
  Other Names: ABI 007; ABI-007; Abraxane; Albumin-bound Paclitaxel; Albumin-Stabilized Nanoparticle Paclitaxel; Nanoparticle Albumin-bound Paclitaxel; Nanoparticle Paclitaxel; Paclitaxel Albumin; paclitaxel albumin-stabilized nanoparticle formulation; Protein-bound Paclitaxel

SUMMARY:
This early phase I trial studies the side effects and feasibility of cryoablation, atezolizumab, and nab-paclitaxel in treating patients with triple negative breast cancer that has spread to nearby tissue or lymph nodes (locally advanced) or has spread to other places in the body (metastatic). Cryosurgery, also known as cryoablation or cryotherapy, kills tumor cells by freezing them. Immunotherapy with monoclonal antibodies, such as atezolizumab, may help the body's immune system attack the cancer, and may interfere with the ability of tumor cells to grow and spread. Drugs used in chemotherapy, such as nab-paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving cryoablation, atezolizumab and nab-paclitaxel may improve response to the disease.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine the safety and feasibility of cryoablation of a primary breast tumor followed by PD-L1 blockade in patients with locally advanced or metastatic triple negative breast cancer (TNBC).

SCONDARY OBJECTIVE:

I. To evaluate the systemic immune response to cryoablation of a primary breast tumor and PD-L1 blockade.

OUTLINE:

Patients undergo cryoablation of the primary tumor over about 1 hour. After 2-3 weeks, patients receive atezolizumab intravenously (IV) on days 1 and 15 and nab-paclitaxel IV on days 1, 8, and 15. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 2-3 weeks post surgery and then periodically thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic PD-L1 positive TNBC (TNBC is defined as estrogen receptor [ER] < 10%, progesterone receptor [PR] < 10%, and HER2 non-amplified; and PD-L1 positive is defined as >= 1%.)
* Presents with primary breast tumor lesion amenable to cryoablation
* Have at least one additional distant lesion feasible for biopsies
* Agreeable to start on atezolizumab and nab-paclitaxel as per standard of care
* Patients with locally advanced disease must be ineligible for curative surgery for any reason, including but not limited to comorbid status precluding surgery due to safety, unresectability, or patient refusal
* Patient may have received prior systemic chemotherapy regimens

Exclusion Criteria:

* History of autoimmune disease
* History of human immunodeficiency virus (HIV)
* Previous immune checkpoint targeting therapies
* No primary breast lesion amenable for cryoablation due to size (greater than 5 cm) or location (proximity of < 0.5 cm to the skin or nipple-areola complex)
* Pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-23 (Actual); Primary Completion 2021-11-17 (Actual); Study Completion 2021-11-17 (Actual)

PRIMARY OUTCOMES:
Safety and Feasibility of cryoablation with systemic atezolizumab/nab-paclitaxel | 5 years
  All adverse events will be reported by grade using frequencies and relative frequencies, and rates will be estimated using a 90% confidence interval obtained using Jeffrey's prior method.

SECONDARY OUTCOMES:
Abscopal response in the distant non-cryoablated site(s) | 5 years
  Will be assessed by using digital spatial profiling. Each immune response will be treated as a continuous variable, and will be summarized using frequencies and relative frequencies. The overall immune response rate will be estimated using a 90% confidence interval obtained using Jeffrey's prior method.
Systemic effector cell and cytokine responses | At baseline, after cryoablation, and after atezolizumab and nab-paclitaxel
  Each immune response will be treated as a continuous variable, and will be summarized using frequencies and relative frequencies. The overall immune response rate will be estimated using a 90% confidence interval obtained using Jeffrey's prior method.
Overall survival | Assessed up to 5 years
  Will be summarized using standard Kaplan-Meier methods. OS defined as Time from cryoablation until death due to any cause or last follow-up
Disease-specific survival | Time from cryoablation until death due to breast cancer or last follow-up, assessed up to 5 years
  Will be summarized using standard Kaplan-Meier methods. OS defined as Time from cryoablation until death due to breast cancer
Progression-free survival | Time from cryoablation to tumor growth as defined by modified Response Evaluation Criteria in Solid Tumors (RECIST) criteria, assessed up to 5 years
  Will be summarized using standard Kaplan-Meier methods.

CONTACTS AND LOCATIONS:
Overall Officials: Emmanuel M Gabriel, Principal Investigator — Mayo Clinic

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials